CLINICAL TRIAL: NCT00804986
Title: A 12-Week,Double-Blind, Placebo-Controlled Trial of LY2428757 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study for Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12134; I1I-MC-GECD (Other: Eli Lilly and Company); CTRI/2009/091/000091 (Registry Identifier: India)
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- 0.5 mg LY2428757 (Experimental): Once weekly, subcutaneous injection of 0.5 milligram (mg) LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: LY2428757
- 2.0 mg LY2428757 (Experimental): Once weekly, subcutaneous injection of 2.0 mg LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: LY2428757
- 6.2 mg LY2428757 (Experimental): Once weekly, subcutaneous injection of 6.2 mg LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: LY2428757
- 12.0 mg LY2428757 (Experimental): Once weekly, subcutaneous injection of 12.0 mg LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: LY2428757
- 17.6 mg LY2428757 (Experimental): Once weekly, subcutaneous injection of 17.6 mg LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: LY2428757
- Placebo (Placebo Comparator): Once weekly, subcutaneous injection of placebo for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2428757 — Once weekly for 12 weeks as a subcutaneous injection.
  Arms: 0.5 mg LY2428757; 12.0 mg LY2428757; 17.6 mg LY2428757; 2.0 mg LY2428757; 6.2 mg LY2428757
Drug: Placebo — 1 of 5 volumes of placebo given once weekly for 12 weeks as a subcutaneous injection.
  Arms: Placebo

SUMMARY:
A multicenter, multinational, randomized,double-blind, placebo-controlled study in patients with Type 2 Diabetes Mellitus (T2DM). Patients with inadequate glycemic control using diet and exercise alone, or in combination with metformin, will be enrolled. The primary objective of this study is to test the hypothesis that LY2428757 given to patients with T2DM inadequately controlled with diet and exercise alone, or metformin monotherapy, produces a significant decrease in the mean hemoglobin A1c (HbA1c) from baseline to endpoint at 12 weeks as compared to placebo. Trial consists of 12 weeks of double-blind treatment and 4-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus for at least 6 months prior to entering the trial.
* Treated with diet and exercise alone or in combination with at least 1000 milligrams (mg)/day of metformin for at least 2 months prior to screening.
* Have a glycosylated fraction of hemoglobin A (HbA1c) value of 7.0% - 10.0% at screening
* Women of child-bearing potential must test negative for pregnancy at screening and agree to abstain from heterosexual intercourse for the duration of the study, or use 2 effective forms of birth control during the study.
* Have a body mass index (BMI) between 25 and 40 kilograms per square meters kg/m^2) at screening
* Stable weight during the 3 months prior to screening.

Exclusion Criteria:

* Use any antidiabetic agent other than metformin during the 2 months prior to screening.
* Have a gastrointestinal disease that significantly impacts gastric emptying or motility or have undergone bariatric surgery.
* Are currently taking prescription or over-the counter medications to promote weight loss.
* Have been previously diagnosed with pancreatitis
* Women who are breastfeeding.
* Have a history of myocardial infarction, unstable angina, coronary artery bypass graft (CABG), percutaneous coronary intervention, transient ischemic attack, stroke or decompensated congestive heart failure in the past 6 months.
* Have poorly controlled hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (60):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bermuda Dunes, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pomona, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waltham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mentor, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vorarlberg
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cooperage
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shivājīnagar
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garza García
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras, Puerto Rico
- Romania (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Satu Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sf Gheorghe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- South Africa (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benoni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempton Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Compostela
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Ukraine (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirovograd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath, Banes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnsley
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5 mg LY2428757: Once weekly, subcutaneous injection of 0.5 mg LY2428757 for 12 weeks. All injections were administered by study site personnel who were blinded to treatment assignment.
Period: Overall Study
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Started | 36 | 43 | 42 | 42 | 43 | 41
Completed | 35 | 35 | 40 | 34 | 34 | 31
Not Completed | 1 | 8 | 2 | 8 | 9 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 3 | 5 | 3
Not completed — Inclusion/Exclusion criteria not met | 0 | 2 | 0 | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo | Total
Number analyzed (Participants) | 36 | 43 | 42 | 42 | 43 | 41 | 247
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.06) | 54.6 (8.33) | 56.4 (8.07) | 55.2 (9.78) | 54.0 (9.45) | 56.3 (9.88) | 55.2 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 24 | 18 | 22 | 24 | 123
  Male | 21 | 23 | 18 | 24 | 21 | 17 | 124
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 4 | 1 | 4 | 1 | 3 | 15
  Asian | 1 | 1 | 3 | 1 | 0 | 1 | 7
  Black or African American | 9 | 6 | 8 | 6 | 10 | 8 | 47
  Native Hawaiian or Pacific Islander | 0 | 1 | 1 | 1 | 0 | 0 | 3
  White | 24 | 31 | 29 | 30 | 32 | 28 | 174
  Multiple Race | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 17 | 12 | 18 | 16 | 19 | 93
  Mexico | 2 | 4 | 1 | 4 | 2 | 4 | 17
  Spain | 0 | 0 | 1 | 1 | 2 | 0 | 4
  Ukraine | 4 | 4 | 9 | 5 | 7 | 5 | 34
  Romania | 4 | 5 | 6 | 5 | 3 | 1 | 24
  Austria | 4 | 2 | 0 | 1 | 0 | 0 | 7
  South Africa | 10 | 8 | 10 | 6 | 8 | 7 | 49
  Germany | 1 | 2 | 3 | 2 | 5 | 4 | 17
  United Kingdom | 0 | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1C (HbA1c) From Baseline to Week 12 Endpoint
Description: LSMean adjusted for baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: Modified intention to treat population, defined as all randomized participants with at least one post-baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 34 | 34 | 39 | 32 | 35 | 32
percentage of glycosylated hemoglobin | -0.60 [-0.87 to -0.34] | -0.80 [-1.05 to -0.55] | -1.24 [-1.49 to -1.00] | -1.41 [-1.67 to -1.15] | -1.37 [-1.62 to -1.11] | -0.13 [-0.39 to 0.13]
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis — p-value represents change from baseline to Week 12 HbA1c for 0.5 mg treatment arm in comparison to placebo with values <0.05 considered to be statistically significant; Mixed effects model: baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -0.47, 95% CI 2-sided [-0.83 to -0.11]
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — p-value represents change from baseline to week 12 HbA1c for 2.0 mg treatment arm in comparison to placebo with values <0.05 considered to be statistically significant; Mixed effects model: baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -0.67, 95% CI 2-sided [-1.02 to -0.31]
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 HbA1c for 6.2 mg treatment arm in comparison to placebo with values <0.05 considered to be statistically significant; Mixed effects model: baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1.11, 95% CI 2-sided [-1.46 to -0.76]
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 HbA1c for 12.0 mg treatment arm in comparison to placebo with values <0.05 considered to be statistically significant; Mixed effects model: baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1.28, 95% CI 2-sided [-1.64 to -0.93]
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 HbA1c for 17.6 mg treatment arm in comparison to placebo with values <0.05 considered to be statistically significant; Mixed effects model: baseline HbA1c, metformin use, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1.24, 95% CI 2-sided [-1.59 to -0.88]

2. Secondary Outcome: Change in Visual Analogue Scales (VAS) For Appetite and Satiety From Baseline to Week 12 Endpoint
Description: The VAS scales for appetite (hunger) and satiety (how full) were recorded on a scale with range of possible scores from 0 to 100 represented in millimeters on a 10 centimeter line. For appetite, participant chooses where they think their appetite lies on a 10 centimeter line between two anchors (0 - not at all hungry and 10 - extremely hungry). For satiety, participant chooses where they think their satiety lies on a 10 centimeter line between two anchors (0 - not at all full and 10 - extremely full). LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 34 | 34 | 38 | 34 | 35 | 34
millimeters (mm)
  Hunger | -2.28 (3.05) | -0.85 (3.03) | -3.76 (2.88) | -0.92 (3.04) | -1.37 (3.00) | -4.22 (3.05)
  How Full | 13.32 (3.53) | 3.04 (3.48) | 5.98 (3.33) | 2.38 (3.50) | 4.41 (3.44) | 10.43 (3.49)
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.655, Mixed Models Analysis — p-value represents change from baseline to Week 12 for hunger, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 1.93
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.436, Mixed Models Analysis — p-value represents change from baseline to Week 12 for hunger, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 3.36
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.914, Mixed Models Analysis — p-value represents change from baseline to Week 12 for hunger, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 0.45
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.446, Mixed Models Analysis — p-value represents change from baseline to Week 12 for hunger, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 3.30
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.508, Mixed Models Analysis — p-value represents change from baseline to Week 12 for hunger, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 2.84
Statistical Analysis 6: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.561, Mixed Models Analysis — p-value represents change from baseline to Week 12 for how full, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = 2.89
Statistical Analysis 7: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.135, Mixed Models Analysis — p-value represents change from baseline to Week 12 for how full, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -7.40
Statistical Analysis 8: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis — p-value represents change from baseline to Week 12 for how full, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -4.45
Statistical Analysis 9: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis — p-value represents change from baseline to Week 12 for how full, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -8.05
Statistical Analysis 10: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.221, Mixed Models Analysis — p-value represents change from baseline to Week 12 for how full, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -6.02

3. Secondary Outcome: Number of Participants With Detectable Antibodies To LY2428757 At Any Time During The Study
Description: Blood samples were collected from all randomized participants to test for the development of antibodies binding to LY2428757. If a participant developed a positive anti-LY2428757 antibody titer, appropriate medical management was to be utilized at the discretion of the sponsor and investigator, if deemed necessary.
Time Frame: baseline through 16 weeks
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 36 | 43 | 42 | 42 | 43 | 41
participants | 1 | 2 | 1 | 3 | 2 | 1

4. Secondary Outcome: Total Average Concentration (Cavg) of LY2428757
Description: Average concentration (Cavg) is calculated as the AUC0-168 (area under the plasma concentration vs. time curve during one dosing interval of 168 hours) divided by 168 hours. The numbers presented reflect the average LY2428757 drug concentration circulating in the body over 168 hours (one dosing interval).
Time Frame: 4 weeks, 6 weeks, 8 weeks, 10 weeks
Population: All randomized participants
Measure: Number; unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 34 | 34 | 39 | 32 | 35 | 32
nanograms per milliliter (ng/mL) | 29.5 | 118 | 453 | 877 | 1290 | 0

5. Secondary Outcome: Change in 7-Point Self-Monitored Glucose From Baseline to Week 12 Endpoint
Description: Self-monitored glucose levels measured at 7 timepoints during the day. Timepoints include: fasting pre-breakfast, 2 hours post breakfast, prior to lunch, 2 hours post lunch, prior to dinner, 2 hours post dinner, and prior to bed. LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 30 | 29 | 36 | 30 | 31 | 29
milligrams per deciliter (mg/dL)
  Fasting | -2.14 [-11.15 to 6.87] | -17.08 [-26.06 to -8.11] | -30.13 [-38.41 to -21.84] | -28.05 [-36.85 to -19.26] | -32.85 [-41.51 to -24.20] | 2.39 [-6.67 to 11.46]
  2 Hours Post Breakfast (n=29, 28, 34,28 30,29) | -7.85 [-23.22 to 7.51] | -32.25 [-47.54 to -16.97] | -45.02 [-59.29 to -30.74] | -45.58 [-60.90 to -30.26] | -53.91 [-68.67 to -39.15] | -2.53 [-17.77 to 12.71]
  Prior to Lunch (n=29, 27, 34, 28, 29, 28) | -6.22 [-19.31 to 6.87] | -7.92 [-21.17 to 5.33] | -25.42 [-37.59 to -13.26] | -22.09 [-35.20 to -8.98] | -26.37 [-39.16 to -13.58] | 13.98 [0.75 to 27.21]
  2 Hours Post Lunch (n=28, 27, 35, 28, 30, 29) | -17.71 [-31.16 to -4.26] | -23.79 [-37.28 to -10.29] | -44.43 [-56.57 to -32.29] | -35.97 [-49.25 to -22.69] | -54.77 [-67.64 to -41.90] | -11.30 [-24.50 to 1.90]
  Prior to Dinner (n=29, 27, 35, 28, 29, 29) | -24.25 [-36.63 to -11.86] | -33.82 [-46.46 to -21.17] | -38.10 [-49.37 to -26.83] | -39.90 [-52.36 to -27.43] | -45.82 [-58.04 to -33.59] | 0.45 [-11.87 to 12.76]
  2 Hours Post Dinner (n=29, 28, 35, 29, 29, 29) | -13.35 [-27.58 to 0.89] | -22.63 [-37.07 to -8.20] | -36.70 [-49.70 to -23.70] | -31.10 [-45.23 to -16.97] | -51.41 [-65.48 to -37.33] | -1.51 [-15.69 to 12.68]
  Prior to Bed (n=27, 23, 33, 25, 29, 25) | -12.33 [-26.37 to 1.70] | -24.08 [-38.94 to -9.23] | -26.48 [-39.23 to -13.72] | -29.05 [-43.33 to -14.78] | -41.48 [-54.74 to -28.21] | 11.69 [-2.82 to 26.19]
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.4848, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -4.54
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -19.48
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -32.52
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -30.45
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -35.25
Statistical Analysis 6: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.6279, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post breakfast glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -5.32
Statistical Analysis 7: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post breakfast glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -29.72
Statistical Analysis 8: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post breakfast glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -42.49
Statistical Analysis 9: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post breakfast glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -43.05
Statistical Analysis 10: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post breakfast glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -51.38
Statistical Analysis 11: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0335, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to lunch glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -20.21
Statistical Analysis 12: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0221, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to lunch glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -21.91
Statistical Analysis 13: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to lunch glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -39.41
Statistical Analysis 14: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to lunch glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -36.07
Statistical Analysis 15: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to lunch glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -40.36
Statistical Analysis 16: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.5030, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post lunch glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -6.41
Statistical Analysis 17: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.1938, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post lunch glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -12.49
Statistical Analysis 18: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post lunch glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -33.13
Statistical Analysis 19: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post lunch glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -24.66
Statistical Analysis 20: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post lunch glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -43.47
Statistical Analysis 21: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0060, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to dinner glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -24.69
Statistical Analysis 22: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to dinner glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -34.26
Statistical Analysis 23: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to dinner glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -38.55
Statistical Analysis 24: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to dinner glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -40.34
Statistical Analysis 25: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to dinner glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -46.26
Statistical Analysis 26: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.2468, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post dinner glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -11.84
Statistical Analysis 27: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0413, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post dinner glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, visit, treatment and visit by treatment interaction as fixed effects; Difference in mean change from baseline = -21.13
Statistical Analysis 28: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post dinner glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -35.19
Statistical Analysis 29: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post dinner glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -29.59
Statistical Analysis 30: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for 2 hours post dinner glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -49.90
Statistical Analysis 31: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0199, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to bed glucose, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -24.02
Statistical Analysis 32: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to bed glucose, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -35.77
Statistical Analysis 33: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to bed glucose, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -38.17
Statistical Analysis 34: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to bed glucose, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -40.74
Statistical Analysis 35: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 for prior to bed glucose, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -53.16

6. Secondary Outcome: Change in Total Glucose Area Under the Curve (AUC) From Baseline to Week 12 Endpoint
Description: An oral glucose tolerance test (OGTT) was used to assess changes in glucose tolerance. The area under the plasma glucose concentration versus time curve was calculated using the linear-trapezoidal method. Area under the curve (AUC) for glucose represents the area that is under the curve of glucose values when they are plotted over time. Larger AUC values represent a greater average glucose value over time. LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per minute per deciliter
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 30 | 28 | 35 | 27 | 32 | 29
milligrams per minute per deciliter | -1370.49 [-3304.81 to 563.83] | -1709.67 [-3710.31 to 290.96] | -5786.59 [-7581.00 to -3992.17] | -6354.83 [-8398.99 to -4310.66] | -8025.33 [-9897.49 to -6153.17] | -238.64 [-2204.37 to 1727.09]
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.4193, Mixed Models Analysis — p-value represents change from baseline to Week 12 total glucose AUC for 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1131.85
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.3026, Mixed Models Analysis — p-value represents change from baseline to Week 12 total glucose AUC for 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1471.04
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 total glucose AUC for 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -5547.95
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 total glucose AUC for 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -6116.19
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value represents change from baseline to Week 12 total glucose AUC for 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -7786.69

7. Secondary Outcome: Change in Insulin Total Area Under the Curve (AUC) From Baseline to Week 12 Endpoint
Description: An oral glucose tolerance test (OGTT) was used to assess changes in insulin secretory response. The area under the insulin concentration versus time curve was calculated using the linear-trapezoidal method. Area under the curve (AUC) for insulin represents the area that is under the curve of insulin values when they are plotted over time. Larger AUC values represent a greater average insulin value over time. LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: picomole per minute per liter
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 23 | 23 | 32 | 23 | 27 | 27
picomole per minute per liter | 3111.25 [-4046.98 to 10269.49] | 3984.37 [-3119.75 to 11088.50] | 12521.89 [6225.80 to 18817.99] | 14179.28 [6829.94 to 21528.62] | 8778.23 [2213.32 to 15343.14] | 3540.52 [-3092.57 to 10173.62]

8. Secondary Outcome: Change in C-peptide Area Under the Curve (AUC) From Baseline to Week 12 Endpoint
Description: An oral glucose tolerance test (OGTT) was used to assess changes in insulin secretory response. The area under the C-peptide concentration versus time curve was calculated using the linear-trapezoidal method. Area under the curve (AUC) for C-peptide represents the area that is under the curve of C-peptide values when they are plotted over time. Larger AUC values represent a greater average C-peptide value over time. LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: picomole per minute per liter
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 29 | 27 | 33 | 27 | 30 | 30
picomole per minute per liter | -683.72 [-27307.99 to 25940.55] | 31434.85 [4250.94 to 58618.75] | 49370.53 [24438.17 to 74302.88] | 46280.14 [18616.52 to 73943.75] | 22012.58 [-3998.13 to 48023.29] | 8714.30 [-17322.91 to 34751.50]

9. Secondary Outcome: Change in Fasting Lipids From Baseline to Week 12 Endpoint
Description: Fasting lipids were measured after overnight fasting of at least 8 hours. Lipids analyzed include triglycerides, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), and total-cholesterol. LSMean adjusted for baseline and treatment.
Time Frame: baseline, 12 weeks
Population: Modified intention to treat population, defined as all randomized participants with at least one post-baseline measurement. The last post-baseline measurement was carried forward if the value at week 12 was missing.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 35 | 40 | 40 | 37 | 41 | 37
millimole per liter (mmol/L)
  Triglycerides (n=35, 40, 40, 37, 41, 37) | -0.15 (0.139) | 0.08 (0.130) | -0.35 (0.130) | -0.31 (0.135) | -0.31 (0.128) | -0.22 (0.135)
  HDL (n=35, 38, 39, 31, 39, 34) | 0.02 (0.034) | -0.03 (0.032) | -0.03 (0.032) | -0.03 (0.036) | 0.02 (0.032) | 0.01 (0.034)
  LDL (n=35, 37, 39, 31, 39, 34) | 0.0 (0.09) | -0.1 (0.09) | -0.1 (0.09) | 0.0 (0.10) | -0.1 (0.09) | 0.1 (0.09)
  Total cholesterol (n=35, 38, 39, 31, 39, 34) | -0.10 (0.104) | -0.01 (0.100) | -0.30 (0.098) | -0.10 (0.112) | -0.25 (0.099) | 0.02 (0.105)
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.693, ANCOVA — p-value represents change from baseline to Week 12 for fasting triglycerides, 0.5 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = 0.08
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.104, ANCOVA — p-value represents change from baseline to Week 12 for fasting triglycerides, 2.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = 0.31
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.506, ANCOVA — p-value represents change from baseline to Week 12 for fasting triglycerides, 6.2 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.13
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.648, ANCOVA — p-value represents change from baseline to Week 12 for fasting triglycerides, 12.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.09
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.647, ANCOVA — p-value represents change from baseline to Week 12 for fasting triglycerides, 17.6 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.09
Statistical Analysis 6: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.781, ANCOVA — p-value represents change from baseline to Week 12 for fasting HDL, 0.5 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = 0.01
Statistical Analysis 7: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.401, ANCOVA — p-value represents change from baseline to Week 12 for fasting HDL, 2.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.04
Statistical Analysis 8: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.464, ANCOVA — p-value represents change from baseline to Week 12 for fasting HDL, 6.2 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.03
Statistical Analysis 9: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.420, ANCOVA — p-value represents change from baseline to Week 12 for fasting HDL, 12.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.04
Statistical Analysis 10: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.762, ANCOVA — p-value represents change from baseline to Week 12 for fasting HDL, 17.6 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = 0.01
Statistical Analysis 11: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.738, ANCOVA — p-value represents change from baseline to Week 12 for fasting LDL, 0.5 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.04
Statistical Analysis 12: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.277, ANCOVA — p-value represents change from baseline to Week 12 for fasting LDL, 2.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.14
Statistical Analysis 13: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.094, ANCOVA — p-value represents change from baseline to Week 12 for fasting LDL, 6.2 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.21
Statistical Analysis 14: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.792, ANCOVA — p-value represents change from baseline to Week 12 for fasting LDL, 12.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.04
Statistical Analysis 15: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.105, ANCOVA — p-value represents change from baseline to Week 12 for fasting LDL, 17.6 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.21
Statistical Analysis 16: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.403, ANCOVA — p-value represents change from baseline to Week 12 for fasting total cholesterol, 0.5 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.12
Statistical Analysis 17: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.799, ANCOVA — p-value represents change from baseline to Week 12 for fasting total cholesterol, 2.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.04
Statistical Analysis 18: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.029, ANCOVA — p-value represents change from baseline to Week 12 for fasting total cholesterol, 6.2 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.32
Statistical Analysis 19: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.439, ANCOVA — p-value represents change from baseline to Week 12 for fasting total cholesterol, 12.0 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.12
Statistical Analysis 20: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.062, ANCOVA — p-value represents change from baseline to Week 12 for fasting total cholesterol, 17.6 mg treatment arm in comparison to placebo; ANCOVA: baseline and treatment; Difference in mean change from baseline = -0.27

10. Secondary Outcome: Change in Fasting Weight From Baseline to Week 12 Endpoint
Description: LSMean adjusted for baseline, treatment, visit, treatment-by-visit interaction.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 35 | 36 | 40 | 36 | 35 | 34
kilograms (kg) | -0.75 [-1.63 to 0.13] | -0.85 [-1.69 to -0.01] | -2.12 [-2.94 to -1.30] | -1.03 [-1.88 to -0.18] | -2.60 [-3.46 to -1.75] | -0.59 [-1.46 to 0.28]
Statistical Analysis 1: Comparison: 0.5 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.8003, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting weight, 0.5 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -0.16
Statistical Analysis 2: Comparison: 2.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.6736, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting weight, 2.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -0.26
Statistical Analysis 3: Comparison: 6.2 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0123, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting weight, 6.2 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -1.53
Statistical Analysis 4: Comparison: 12.0 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.4771, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting weight, 12.0 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -0.44
Statistical Analysis 5: Comparison: 17.6 mg LY2428757 vs Placebo; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — p-value represents change from baseline to Week 12 for fasting weight, 17.6 mg treatment arm in comparison to placebo; Mixed effects model: baseline, treatment, visit, treatment-by-visit interaction; Difference in mean change from baseline = -2.01

11. Secondary Outcome: Change in Impact of Weight on Quality of Life - Lite (IWQoL-Lite) Average Score From Baseline to Week 12 Endpoint
Description: Impact of Weight on Quality of Life (IWQoL) - Lite Version consists of 31 items from 5 subscales: physical functioning, self-esteem, sexual life, public distress, and work as well as a total score. Individual item scoring ranges from 0 (never true) to 4 (always true) with total score range from 0 to 124. Higher scores on the subscales and total score correspond with lower levels of functioning or greater negative effect. LSMean adjusted for baseline, baseline HbA1c (less than 8.5% versus greater than or equal to 8.5%), metformin use, treatment.
Time Frame: baseline, 12 weeks
Population: Modified intention to treat population, defined as all randomized participants with at least one post-baseline measurement, last observation carried forward (LOCF) up to visit 9 (week 12)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 35 | 39 | 40 | 38 | 40 | 37
units on a scale | 0.2 (0.22) | -0.1 (0.20) | 0.3 (0.21) | 0.2 (0.21) | 0.1 (0.21) | 0.2 (0.21)

12. Secondary Outcome: Change in Diabetes Symptom Checklist-Revised (DSC-R) Average Score From Baseline to Week 12 Endpoint
Description: DSC-R assesses the presence and perceived burden of diabetes-related symptoms using the following subscales: hypoglycemic, hyperglycemic, psychological, cardiovascular, neurological, ophthalmological. Participants evaluate symptoms based on a 5-point Likert-type scale, ranging from 1=not at all troublesome to 5=extremely troublesome. Higher scores indicated greater severity of symptoms within a domain, or poorer perceived health, respectively. LSMean adjusted for baseline, baseline HbA1c (less than 8.5% versus greater than or equal to 8.5%), metformin use, treatment.
Time Frame: baseline, 12 weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 35 | 39 | 40 | 37 | 40 | 38
units on a scale | -0.3 (0.30) | -0.1 (0.28) | -0.9 (0.28) | -0.4 (0.29) | -0.3 (0.29) | -0.7 (0.28)

13. Secondary Outcome: Change in European Quality of Life (EuroQol)- Visual Analog Scale From Baseline to Week 12 Endpoint
Description: Participant chooses where they think their current health state lies on a 10 centimeter line between two anchors (0 - worst imaginable health state and 10 - best imaginable health state). The possible range of scores is 0 to 100 and represents millimeters on the 10 centimeter line. A higher score is associated with better health state. LSMean adjusted for baseline, baseline HbA1c (less than 8.5% versus greater than or equal to 8.5%), metformin use, treatment.
Time Frame: baseline, 12 weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 35 | 39 | 40 | 38 | 40 | 37
millimeters | 6.9 (2.59) | 6.2 (2.33) | 6.0 (2.41) | 6.0 (2.46) | 7.1 (2.47) | 2.7 (2.48)

14. Secondary Outcome: Percent of Participants Domain Scores Indicating No Problems on European Quality of Life (EuroQol) at Baseline and Week 12 Endpoint
Description: The EuroQoL Questionnaire - 5 Dimension (EQ-5D) is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 is generated for each domain. For each participant, the outcome rating on the 5 domains will be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the participant.
Time Frame: Baseline, 12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Number analyzed (Participants) | 36 | 42 | 42 | 39 | 42 | 40
percentage of participants
  Mobility-Baseline | 88.9 | 73.8 | 76.2 | 84.6 | 81.0 | 75.0
  Mobility-Endpoint | 94.3 | 77.8 | 90.0 | 77.8 | 88.6 | 85.3
  Self Care-Baseline | 97.2 | 97.6 | 90.5 | 94.9 | 95.2 | 97.5
  Self Care- Endpoint | 94.3 | 97.2 | 100.0 | 94.4 | 100.0 | 97.1
  Usual Activities- Baseline | 80.6 | 81.0 | 83.3 | 87.2 | 81.0 | 75.0
  Usual Activities- Endpoint | 91.4 | 88.9 | 90.0 | 91.7 | 97.1 | 88.2
  Pain/Discomfort- Baseline | 61.1 | 59.5 | 54.8 | 59.0 | 54.8 | 52.5
  Pain/Discomfort- Endpoint | 60.0 | 52.8 | 70.0 | 63.9 | 71.4 | 61.8
  Anxiety/Depression- Baseline | 66.7 | 64.3 | 73.8 | 74.4 | 66.7 | 70.0
  Anxiety/Depression- Endpoint | 68.6 | 69.4 | 87.5 | 77.8 | 74.3 | 70.6

ADVERSE EVENTS:
Description: The safety population includes all randomized participants who received at least one administration of study medication.
Arm/Group | 0.5 mg LY2428757 | 2.0 mg LY2428757 | 6.2 mg LY2428757 | 12.0 mg LY2428757 | 17.6 mg LY2428757 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/36 | 4/42 | 1/42 | 1/41 | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 19/36 | 25/42 | 26/42 | 24/41 | 28/43 | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg LY2428757 (N=36) | 2.0 mg LY2428757 (N=42) | 6.2 mg LY2428757 (N=42) | 12.0 mg LY2428757 (N=41) | 17.6 mg LY2428757 (N=43) | Placebo (N=40)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg LY2428757 (N=36) | 2.0 mg LY2428757 (N=42) | 6.2 mg LY2428757 (N=42) | 12.0 mg LY2428757 (N=41) | 17.6 mg LY2428757 (N=43) | Placebo (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (7) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (7) | 7 (9) | 3 (4) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5) | 6 (9) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 6 (6) | 9 (21) | 13 (18) | 16 (29) | 6 (6)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 7 (12) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Protein urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (5) | 2 (3) | 5 (5) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days